CLINICAL TRIAL: NCT02085824
Title: Comparison of Blood Loss Following Total Hip Arthroplasty With the Use of Three Thromboprophylactic Regimes: Dabigatran, Enoxaparin and Rivaroxaban.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre of Postgraduate Medical Education (Other)
Responsible Party: Principal Investigator, Marcin Wasko MD PhD, Dr Marcin Wasko MD PhD, Centre of Postgraduate Medical Education
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CPX-2012
Record Dates: First submitted 2014-03-07; First posted 2014-03-13 (Estimated); Last update posted 2014-03-14 (Estimated); Status verified 2014-03

CONDITIONS: Hip Osteoarthritis; Blood Loss
MeSH Terms: conditions — Osteoarthritis, Hip; Hemorrhage | interventions — Enoxaparin; Rivaroxaban; Dabigatran

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- enoxaparin (Experimental): enoxaparin 40mg 1x1 s.c. daily, once preoperatively and then daily for 28 days
  Interventions: Drug: Enoxaparin
- rivaroxaban (Experimental): rivaroxaban 10 mg 1x1 p.o. daily for 28 days after the surgery
  Interventions: Drug: rivaroxaban
- dabigatran (Experimental): dabigatran 110 mg 1x1 p.o. postoperatively and then 1x2 p.o. for 27 days after the surgery
  Interventions: Drug: dabigatran

INTERVENTIONS:
Drug: Enoxaparin
  Arms: enoxaparin
Drug: rivaroxaban
  Arms: rivaroxaban
Drug: dabigatran
  Arms: dabigatran

SUMMARY:
The purpose of this study is to determine which of the following drugs: enoxaparin, dabigatran and rivaroxaban causes least blood loss after total hip replacement (THR).

ELIGIBILITY:
Inclusion Criteria:

* primary, end-stage hip osteoarthritis requiring total hip arthroplasty

Exclusion Criteria:

* inflammatory arthropathies
* liver disorders
* neoplastic conditions
* clotting disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-07; Primary Completion 2014-04 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Total blood loss by the 3rd postoperative day | 3rd day postoperatively
  Measured for each individual. Measured according to the formula described by Nadler, Hidalgo and Bloch (Prediction of blood volume in normal human adults. Surgery 1962;51:224-32).

SECONDARY OUTCOMES:
Drop in the haemoglobin value between 3rd day postop and preoperative | 3rd day postopertively
  Difference between haemoglobin on the 3rd postopertive day and day before operation
Wound healing disturbances according to the definition of Centers for Disease Control and Prevention | 3 months postoperatively
  Wound healing disturbances - diagnosis to be made according to the definition of Centers for Disease Control and Prevention (Mangram, Horan, Pearson, Silver and Jarvis. Guideline for prevention of surgical site infection, 1999. Hospital Infection Control Practices Advisory Committee. Infect Control Hosp Epidemiol. 1999 Apr;20(4):250-78)

CONTACTS AND LOCATIONS:
Overall Officials: Marcin K Wasko, M.D., Ph.D., Principal Investigator — The Medical Centre of Postgraduate Education, Department of Orthopaedics and Inflammatory Disorders of Locomotor System
Locations (1):
- Prof. A. Gruca Teaching Hospital, The Medical Centre of Postgraduate Education, Otwock, Woj. Mazowieckie, Poland